CLINICAL TRIAL: NCT02104427
Title: A Phase II, Open-Label Study to Evaluate the Hematopoietic Stem Cell Mobilization of TG-0054 Combined With G-CSF in Patients With Multiple Myeloma, Non-Hodgkin Lymphoma or Hodgkin Disease
Brief Title: PD and Safety of TG-0054 Combined With G-CSF in Multiple Myeloma, Non-Hodgkin Lymphoma and Hodgkin Disease Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GPCR Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TG-0054-04
Record Dates: First submitted 2014-03-26; First posted 2014-04-04 (Estimated); Results first posted 2017-12-13 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Multiple Myeloma; Non-Hodgkin Lymphoma; Hodgkin Disease
MeSH Terms: conditions — Multiple Myeloma; Lymphoma, Non-Hodgkin; Hodgkin Disease | interventions — Granulocyte Colony-Stimulating Factor

ARMS (1):
- TG-0054 combined with G-CSF (Experimental): 1. G-CSF: 10 μg/kg/day, administrated via SC injections from Day 1 to Day 8; 2. TG-0054: 3.14 mg/kg, administrated via 15-min IV infusion from Day 5 to Day 9 as needed to reach the target collection goal
  Interventions: Drug: TG-0054 combined with G-CSF

INTERVENTIONS:
Drug: TG-0054 combined with G-CSF

SUMMARY:
This is a phase II study to evaluate the efficacy and safety of TG-0054 combined with G-CSF in mobilizing hematopoietic stem cells in patients with multiple myeloma, non-Hodgkin lymphoma or Hodgkin disease.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 to 75 years of age inclusive;
* Patients with confirmed pathology diagnosis of MM, NHL or HD;
* Potential candidate for autologous stem cell transplantation at Investigator's discretion;
* > 4 weeks since last cycle of chemotherapy prior to the study drug administration;
* Total dose of melphalan received ≦ 200 mg in the most recent chemotherapy treatment;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
* Recovered from all acute toxic effects of prior chemotherapy at Investigator's discretion;
* White blood cell (WBC) count ≧ 3.0*10^9/L on screening laboratory assessments;
* Absolute neutrophil count ≧ 1.5*10^9/L on screening laboratory assessments;
* Platelet count ≧ 100*10^9/L on screening laboratory assessments;
* Serum creatinine ≦ 2.2 mg/dL on screening laboratory assessments;
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and total bilirubin < 2 x upper limit of normal (ULN) on screening laboratory assessments;
* Negative for human immunodeficiency virus (HIV);
* Adequate cardiac and pulmonary function to undergo leukapheresis at Investigator's discretion;
* For females, one of the following criteria must be fulfilled:

  1. At least one year post-menopausal, or
  2. Surgically sterile, or
  3. Willing to use a double-barrier method [intrauterine device (IUD) plus condom, spermicidal gel plus condom] of contraception from study Day 1 until 28 days after the last dose of TG-0054;
* Males must be willing to use a reliable form of contraception (use of a condom or a partner fulfilling the above criteria) from study Day 1 until 28 days after the last dose of TG-0054;
* Able to provide the signed informed consent.

Exclusion Criteria:

* Received radiation therapy to the pelvis;
* Received > 6 cycles of lenalidomide;
* Evidence of bone marrow involvement of lymphoma in NHL patients;
* Failed previous stem cell collection [failed to collect 2.0*10^6 CD34+ cells/kg within 4 leukapheresis sessions after receiving granulocyte colony-stimulating factor (G-CSF)];
* Patients who have undergone previous stem cell transplantation procedure;
* Received G-CSF within 2 weeks prior to the study drug administration;
* History of other cancer within the past 5 years excluding MM, NHL, HD, basal cell or squamous cell carcinoma of the skin;
* History of other hematologic disorders including bleeding or thromboembolic disease being treated with anti-coagulant;
* History of poor and uncontrollable cardiovascular or pulmonary disease such as myocardial infarction, cardiac arrhythmias, transient ischemic attack, stroke or Chronic Obstructive Pulmonary Disease (COPD) patients hospitalized more than two times a year due to underlying disease;
* Diagnosis of sickle cell anemia or documented sickle cell trait;
* Patients with proliferative retinopathy;
* Uncontrollable malignancy with MM, NHL or HD, or carcinomatous meningitis, at Investigator's discretion;
* Any infection required antibiotic treatment or unexplained fever above 38 °C within 3 days prior to dosing;
* Pregnant or breast-feeding;
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious disease) illness must not be enrolled into this study;
* Received any other investigational drug within 1 month before entering the study;
* Received prior treatment with TG-0054 but withdrew early from this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-02; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael M Schuster, MD, Principal Investigator — Stony Brook University Hospital
Locations (2):
- United States (2):
  - Stony Brook University Hospital, Stony Brook, New York
  - Tennessee Oncology, PLLC, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TG-0054 Combined With G-CSF
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | TG-0054 Combined With G-CSF
Number analyzed (Participants) | 12
Age, Continuous [Mean (Full Range); unit: years] | 58 [41 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 2
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Weight [Mean (Full Range); unit: kg] | 82.4 [54.6 to 114.0]
BMI [Mean (Full Range); unit: kg/m^2] | 29.3 [21.9 to 37.1]

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients From Whom a Total Number of CD34+ Cells ≥5.0 x 10^6 Cells/kg Was Collected Within the First 4 Leukapheresis Sessions
Description: The primary efficacy endpoint was the proportion of patients from whom a total number of CD34+ cells ≥5.0 x 10^6 cells/kg was collected within the first 4 leukapheresis sessions. For the primary efficacy endpoint, each patient's CD34+ cell number was calculated as the sum of CD34+ cell numbers collected from (up to) the first 4 leukapheresis sessions.
Time Frame: Day 5 to Day 8
Population: There were total 9 MM patients and 3 NHL or HD patients . A MM patient was treated with Revlimid, Following 2 leukapheresis sessions, a cumulative total of 0.18 x 10^6 cells/kg were collected. PI and Medical Monitor didn't feel that further leukapheresis sessions would achieve more cells, so the patient didn't have additional sessions.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Groups:
- Within 1 Leukapheresis Session: Cumulative CD34+ cell counts ≥5.0 x 10^6 cells/kg within 1 leukapheresis session
- Within 2 Leukapheresis Sessions: Cumulative CD34+ cell counts ≥5.0 x 10^6 cells/kg within 2 leukapheresis session
- Within 3 Leukapheresis Sessions: Cumulative CD34+ cell counts ≥5.0 x 10^6 cells/kg within 3 leukapheresis session
- Within 4 Leukapheresis Sessions: Cumulative CD34+ cell counts ≥5.0 x 10^6 cells/kg within 4 leukapheresis session
Arm/Group | Within 1 Leukapheresis Session | Within 2 Leukapheresis Sessions | Within 3 Leukapheresis Sessions | Within 4 Leukapheresis Sessions
Number analyzed (Participants) | 12 | 12 | 12 | 12
Proportion of participants
  Overall | 0.50000 [0.2109 to 0.7891] | 0.9167 [0.6152 to 0.9979] | 0.9167 [0.6152 to 0.9979] | 0.9167 [0.6152 to 0.9979]
  Multiple Myeloma: number analyzed (Participants) | 9 | 9 | 9 | 9
  Multiple Myeloma | 0.6667 [0.2993 to 0.9251] | 0.8889 [0.5175 to 0.9972] | 0.8889 [0.5175 to 0.9972] | 0.8889 [0.5175 to 0.9972]
  Non-Hodgkin Lymphoma or Hodgkin Disease: number analyzed (Participants) | 3 | 3 | 3 | 3
  Non-Hodgkin Lymphoma or Hodgkin Disease | 0.0000 [0.0000 to 0.0000] | 1.0000 [0.2924 to 1.0000] | 1.0000 [0.2924 to 1.0000] | 1.0000 [0.2924 to 1.0000]

2. Secondary Outcome: Proportion of Patients From Whom a Total Number of CD34+ Cells ≥2.5 x 10^6 Cells/kg Was Collected Within the First 4 Leukapheresis Sessions
Description: The secondary efficacy endpoint was the proportion of patients from whom a total number of CD34+ cells ≥2.5 x 10^6 cells/kg was collected within the first 4 leukapheresis sessions. Each patient's CD34+ cell number was calculated as the sum of CD34+ cell numbers collected from (up to) the first 4 leukapheresis sessions.
Time Frame: Day 5 to Day 8
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Proportion of patients
Groups:
- Within 1 Leukapheresis Session: Cumulative CD34+ cell counts ≥2.5 x 10^6 cells/kg within 1 leukapheresis session
- Within 2 Leukapheresis Sessions: Cumulative CD34+ cell counts ≥2.5 x 10^6 cells/kg within 2 leukapheresis session
- Within 3 Leukapheresis Sessions: Cumulative CD34+ cell counts ≥2.5 x 10^6 cells/kg within 3 leukapheresis session
Arm/Group | Within 1 Leukapheresis Session | Within 2 Leukapheresis Sessions | Within 3 Leukapheresis Sessions | Within 4 Leukapheresis Sessions
Number analyzed (Participants) | 12 | 12 | 12 | 12
Proportion of patients
  Overall | 0.9167 [0.6152 to 0.9979] | 0.9167 [0.6152 to 0.9979] | 0.9167 [0.6152 to 0.9979] | 0.9167 [0.6152 to 0.9979]
  Multiple Myeloma: number analyzed (Participants) | 9 | 9 | 9 | 9
  Multiple Myeloma | 0.8889 [0.5175 to 0.9972] | 0.8889 [0.5175 to 0.9972] | 0.8889 [0.5175 to 0.9972] | 0.8889 [0.5175 to 0.9972]
  Non-Hodgkin Lymphoma or Hodgkin Disease: number analyzed (Participants) | 3 | 3 | 3 | 3
  Non-Hodgkin Lymphoma or Hodgkin Disease | 1.0000 [0.2924 to 1.0000] | 1.0000 [0.2924 to 1.0000] | 1.0000 [0.2924 to 1.0000] | 1.0000 [0.2924 to 1.0000]

3. Secondary Outcome: Proportion of Patients Who Mobilized the Targeted Total Number of CD34+ Cells (≥6.0 x 10^6 Cells/kg) Within 5 Leukapheresis Sessions
Description: The secondary efficacy endpoint was the proportion of patients from whom a total number of CD34+ cells ≥6.0 x 10^6 cells/kg was collected within 5 leukapheresis sessions. Each patient's CD34+ cell number was calculated as the sum of CD34+ cell numbers collected from (up to) 5 leukapheresis sessions.
Time Frame: Day 5 to Day 9
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Proportion of patients
Groups:
- Within 1 Leukapheresis Session: Cumulative CD34+ cell counts ≥6.0 x 10^6 cells/kg within 1 leukapheresis session
- Within 2 Leukapheresis Sessions: Cumulative CD34+ cell counts ≥6.0 x 10^6 cells/kg within 2 leukapheresis session
- Within 3 Leukapheresis Sessions: Cumulative CD34+ cell counts ≥6.0 x 10^6 cells/kg within 3 leukapheresis session
- Within 4 Leukapheresis Sessions: Cumulative CD34+ cell counts ≥6.0 x 10^6 cells/kg within 4 leukapheresis session
- Within 5 Leukapheresis Sessions: Cumulative CD34+ cell counts ≥6.0 x 10^6 cells/kg within 5 leukapheresis session
Arm/Group | Within 1 Leukapheresis Session | Within 2 Leukapheresis Sessions | Within 3 Leukapheresis Sessions | Within 4 Leukapheresis Sessions | Within 5 Leukapheresis Sessions
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12
Proportion of patients
  Overall | 0.5000 [0.2109 to 0.7891] | 0.6667 [0.3489 to 0.9008] | 0.6667 [0.3489 to 0.9008] | 0.6667 [0.3489 to 0.9008] | 0.6667 [0.3489 to 0.9008]
  Multiple myeloma: number analyzed (Participants) | 9 | 9 | 9 | 9 | 9
  Multiple myeloma | 0.6667 [0.2993 to 0.9251] | 0.8889 [0.5175 to 0.9972] | 0.8889 [0.5175 to 0.9972] | 0.8889 [0.5175 to 0.9972] | 0.8889 [0.5175 to 0.9972]
  Non-Hodgkin Lymphoma or Hodgkin Disease: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3
  Non-Hodgkin Lymphoma or Hodgkin Disease | 0.0000 [0.0000 to 0.0000] | 0.0000 [0.0000 to 0.0000] | 0.0000 [0.0000 to 0.0000] | 0.0000 [0.0000 to 0.0000] | 0.0000 [0.0000 to 0.0000]

4. Secondary Outcome: the Pharmacodynamics (PD) Following Treatment With TG-0054 When Combined With G-CSF
Description: determine circulating CD34+ cell counts in peripheral blood
Time Frame: Day 5 (1st leukapheresis session) to Day 6 (2nd leukapheresis session)
Population: There were 5 patients who achived target number of CD34+ cells (>=5.0*10^6 cells/kg) within two leukapheresis sessions and therefore didn't undergo addtional sessions. Among 7 patients who undergone 6 sessions, there were 1 patient didn't collect blood sample at 4h, 6h post-infusion and post-leukapheresis, and 1 patient 6h post-infusion not done.
Measure: Median (Full Range); unit: cells/µL
Groups:
- Pre-dose: Circulating CD34+ Cell Count (cells/µL) in Peripheral Blood at Pre-dose timepoint
- 4h Post-infusion: Circulating CD34+ Cell Count (cells/µL) in Peripheral Blood at 4h post-infusion timepoint
- 6h Post-infusion: Circulating CD34+ Cell Count (cells/µL) in Peripheral Blood at 6h post-infusion timepoint
- Pre-leukapheresis: Circulating CD34+ Cell Count (cells/µL) in Peripheral Blood at Pre-leukapheresis timepoint
- Post-leukapheresis: Circulating CD34+ Cell Count (cells/µL) in Peripheral Blood at Post-leukapheresis timepoint
Arm/Group | Pre-dose | 4h Post-infusion | 6h Post-infusion | Pre-leukapheresis | Post-leukapheresis
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12
cells/µL
  Day 5 (1st leukapheresis session) | 32.50 [1.00 to 123.00] | 43.50 [0.00 to 141.00] | 42.00 [1.00 to 122.00] | 60.50 [1.00 to 206.00] | 35.50 [3.00 to 119.00]
  Day 6 (2nd leukapheresis session): number analyzed (Participants) | 7 | 6 | 5 | 7 | 6
  Day 6 (2nd leukapheresis session) | 16.00 [1.00 to 59.50] | 28.00 [14.00 to 45.00] | 20.00 [0.00 to 45.00] | 34.00 [2.00 to 70.00] | 21.00 [16.00 to 45.00]

ADVERSE EVENTS:
Groups:
- 10 µg/kg/Day G-CSF Alone: Days 1 through 4
- 10 µg/kg/Day G-CSF + 3.14 mg/kg TG-0054: Day 5 until end of study
Arm/Group | 10 µg/kg/Day G-CSF Alone | 10 µg/kg/Day G-CSF + 3.14 mg/kg TG-0054 | Overall
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 2/12 | 6/12 | 7/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10 µg/kg/Day G-CSF Alone (N=12) | 10 µg/kg/Day G-CSF + 3.14 mg/kg TG-0054 (N=12) | Overall (N=12)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days